CLINICAL TRIAL: NCT04664790
Title: Hyperbaric Oxygen Therapy vs. Cognitive Training for Fetal Alcohol Spectrum Disorder; A Prospective, Randomized Clinical Trial
Brief Title: Hyperbaric Oxygen Therapy Compared to Cognitive Training in FASD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 275-20-ASF
Record Dates: First submitted 2020-11-24; First posted 2020-12-11 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: FASD
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Hyperbaric Oxygenation; Cognitive Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric Oxygen (Active Comparator): 60 daily hyperbaric oxygen treatment sessions will be administrated 5 days per week.
  Interventions: Device: Hyperbaric Oxygen
- Cognitive training (Active Comparator): Neuropsychologist guided cognitive training.
  Interventions: Behavioral: Cognitive training

INTERVENTIONS:
Device: Hyperbaric Oxygen — Each session will include exposure of 90 minutes to 100% at 2 ATA, with 5 minutes air breaks every 20 minutes
  Arms: Hyperbaric Oxygen
Behavioral: Cognitive training — Neuropsychologist guided BrainHQ training
  Arms: Cognitive training

SUMMARY:
Fetal Alcohol Spectrum Disorder (FASD) describes a wide range of adverse physical, behavioral and cognitive effects resulting from prenatal alcohol exposure (PAE) during embryonic and fetal development. A number of clinical studies have presented evidence regarding the physiological effects of HBOT on metabolically dysfunctional brain regions that might be related to FASD. The aim of the study is to compare the effect of HBOT vs. neurocognitive training on neurobehavioral function in FASD.

DETAILED DESCRIPTION:
Fetal Alcohol Spectrum Disorder (FASD) describes a wide range of adverse physical, behavioral and cognitive effects resulting from prenatal alcohol exposure (PAE) during embryonic and fetal development. Currently individuals afflicted by FASD are treated symptomatically for ADHD and different forms of disruptive behavior. However, these approaches have not succeeded in improving the long-term clinical outcome [1].

A number of clinical studies have presented evidence regarding the physiological effects of hyperbaric oxygen therapy (HBOT) on metabolically dysfunctional brain regions that might be related to FASD [2-5]. Case studies conducted using HBOT suggested a potential safe and efficient treatment for FESD [6-7]. The aim of the study is to compare the effect of HBOT vs. neurocognitive training on neurobehavioral function in FASD.

The study is designed as a prospective randomized, two active arm trial. After enrolment, eligible participants will be randomized with equal probability into one of two arms: HBOT or cognitive training arm. The evaluation procedure will be performed twice, at baseline and 1-3 weeks after the last treatment session, and includes cognitive tests, FASD relegated questionnaires, and anatomical and functional brain imaging (MRI and SPECT). The study is designed as an intention to treat trial, and thus, patients will be included in the analysis if they completed at least one HBOT/cognitive training session, and attained post treatment study analysis.

The HBOT protocol will be administrated in a multi-place chamber. The protocol comprised of 60 daily sessions, 5 sessions per week within a three month period. Each session includes breathing 100% oxygen by mask at 2ATA for 90 minutes with 5-minute air breaks every 20 minutes.

The cognitive training protocol contains a neuropsychologist guided BrainHQ training program. This is a 3 months program that includes 30 minutes sessions at least 3 times per week.

ELIGIBILITY:
Inclusion Criteria:

* Subject willing and able to sign an informed consent
* Age 18 years and older
* Diagnosed with FASD by an Israeli expert
* Failure to improve after at least one line of conventional therapy
* Stable psychological and pharmacological treatment for over three months prior to inclusion

Exclusion Criteria:

* Inability to attend scheduled clinic visits and/or comply with the study protocol
* History of other brain pathologies
* Active malignancy
* Serious suicidal ideation
* Severe or unstable physical disorders at baseline
* History of HBOT for any reason prior to study enrollment
* Chest pathology incompatible with pressure changes (including active asthma)
* Inner ear disease
* Contraindications for MRI or inability to perform an awake brain MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive health assessment (NeuroTrax) | baseline, 3 months
  Memory, attention and information process will be evaluated using the NeuroTrax computerized cognitive evaluation battery.
Executive functions and self-regulation in everyday environment | baseline, 3 months
  Evaluated using the Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) self-reported questionnaire

SECONDARY OUTCOMES:
Brain perfusion | baseline, 3 months
  Cerebral blood volume and flow will be measured using perfusion MRI protocol Dynamic susceptibility contrast (DSC).
Brain microstructure - (MD) | baseline, 3 months
  Mean diffusivity (MD) will be evaluated using diffusion tensor imaging (DTI) MRI protocol.
Brain microstructure - (FA) | baseline, 3 months
  Fractional anisotropy (FA) will be evaluated using diffusion tensor imaging (DTI) MRI protocol.
Brain function imaging | baseline, 3 months
  Resting state fMRI (rsfMRI), and task based fmri will evaluate brain function during a working memory task.
Metabolic Brain function imaging | baseline, 3 months
  Brain Single photon emission computed tomography (SPECT) will be conducted using Tc-99m-ECD.
Depression anxiety and stress | baseline, 3 months, 6 months
  Evaluated using the Depression Anxiety Stress Scale Test (DASS 21) self-report instrument.
Interpersonal Reactive Index (IRI) | baseline, 3 months, 6 months
  The IRI questionnaire will be used to evaluate cognitive and affective aspects of empathic abilities.
Difficulties in Emotion Regulation Scale (DERS) | baseline, 3 months, 6 months
  The DERS questionnaire is a multidimensional self-report measure of emotion regulation
Mental Health Continuum (MHC-SF) | baseline, 3 months, 6 months
  The MHC-SF questionnaire will be used to assess three components of well-being: emotional, social, and psychological and conduct categorical diagnosis of positive mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Background] Goodlett CR, Horn KH. Mechanisms of alcohol-induced damage to the developing nervous system. Alcohol Res Health. 2001;25(3):175-84. PMID 11810955
- [Background] Efrati S, Ben-Jacob E. Reflections on the neurotherapeutic effects of hyperbaric oxygen. Expert Rev Neurother. 2014 Mar;14(3):233-6. doi: 10.1586/14737175.2014.884928. Epub 2014 Jan 29. PMID 24471697
- [Background] Efrati S, Fishlev G, Bechor Y, Volkov O, Bergan J, Kliakhandler K, Kamiager I, Gal N, Friedman M, Ben-Jacob E, Golan H. Hyperbaric oxygen induces late neuroplasticity in post stroke patients--randomized, prospective trial. PLoS One. 2013;8(1):e53716. doi: 10.1371/journal.pone.0053716. Epub 2013 Jan 15. PMID 23335971
- [Background] Hadanny A, Bechor Y, Catalogna M, Daphna-Tekoah S, Sigal T, Cohenpour M, Lev-Wiesel R, Efrati S. Hyperbaric Oxygen Therapy Can Induce Neuroplasticity and Significant Clinical Improvement in Patients Suffering From Fibromyalgia With a History of Childhood Sexual Abuse-Randomized Controlled Trial. Front Psychol. 2018 Dec 17;9:2495. doi: 10.3389/fpsyg.2018.02495. eCollection 2018. PMID 30618929
- [Background] Hadanny A, Rittblat M, Bitterman M, May-Raz I, Suzin G, Boussi-Gross R, Zemel Y, Bechor Y, Catalogna M, Efrati S. Hyperbaric oxygen therapy improves neurocognitive functions of post-stroke patients - a retrospective analysis. Restor Neurol Neurosci. 2020;38(1):93-107. doi: 10.3233/RNN-190959. PMID 31985478
- [Background] Stoller KP. Quantification of neurocognitive changes before, during, and after hyperbaric oxygen therapy in a case of fetal alcohol syndrome. Pediatrics. 2005 Oct;116(4):e586-91. doi: 10.1542/peds.2004-2851. Epub 2005 Sep 15. PMID 16166387
- [Background] Koren G, Golan C, Suzin G, Berkovich M, Efrati S. Effects of Hyperbaric Oxygen Therapy on Brain Perfusion, Cognition and Behavior in Fetal Alcohol Spectrum Disorder-A Case Study. Alcohol Alcohol. 2019 Mar 1;54(2):177-179. doi: 10.1093/alcalc/agz009. PMID 30801636